CLINICAL TRIAL: NCT02946827
Title: The Efficacy of a Low FODMAPs (Fermentable Oligo- di- and Monosaccharides and Polyols) Diet in Celiac Patients With Persistent Gastrointestinal Symptoms
Brief Title: A Low FODMAPs Diet in Celiac Patients With Persistent Gastrointestinal Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Leda Roncoroni, BS PhD, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/464
Record Dates: First submitted 2016-10-18; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Celiac Disease
Keywords: FODMAPs diet; micro-macro nutrients intake; IBS (Irritable Bowel Syndrome)
MeSH Terms: conditions — Celiac Disease; Irritable Bowel Syndrome | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low FODMAPs /balanced gluten free diet (Experimental): An expert in nutrition will give a balanced gluten free diet to patients, low in FODMAPs foods.
  Interventions: Dietary Supplement: Balanced low FODMAPs /gluten free diet
- Balanced gluten free diet (Active Comparator): An expert in nutrition will give a balanced gluten free diet to patients.
  Interventions: Dietary Supplement: Balanced gluten free diet

INTERVENTIONS:
Dietary Supplement: Balanced low FODMAPs /gluten free diet
  Arms: Low FODMAPs /balanced gluten free diet
Dietary Supplement: Balanced gluten free diet
  Arms: Balanced gluten free diet

SUMMARY:
FODMAPS (fructose, oligosaccharides, monosaccharides, disaccharides and polyols) are characterised as fermentable but poorly absorbed carbohydrates which enter the colon and are utilised by colonic bacteria. During fasting colonic nutrients are scarce but ingesting FODMAPS causes a rapid increase in carbohydrate which can overwhelm the microbiota's ability to utilise substrate. The excess reducing equivalents will generate hydrogen or methane. The principal symptoms are diarrhoea and abdominal distension. Patients with irritable bowel syndrome appear to benefit by restricting intake, possibly because they are hypersensitive to intestinal distension.

The focus of the study is to evaluate if in celiac patients with persistent abdominal symptoms and with a correct gluten free diet, a low FODMAPs diet can improve their symptoms. Moreover the study would like to observe if a dietary restriction in FODMAPs carries the risk of nutritional inadequacy.

ELIGIBILITY:
Inclusion Criteria:

* Celiac patients assessed through positive serology and histology
* functional patients according IBS Roma III criteria
* subjects with VAS>5

Exclusion Criteria:

* refractory celiac disease
* disaccharide intolerance (fructose an lactose breath test)
* abdominal surgery
* comorbidity
* patients recruited in other clinical trials
* positive patients at lactulose breath test (SIBO)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of VAS (psychometric response scale level continuous line between two end-points 0-10) values of globel well-being in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients in balanced gluten free diet. | 21 days

SECONDARY OUTCOMES:
Improvement of VAS values of IBS symptoms in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients undergoing only a balanced gluten free diet. | 21 days
  Evaluated IBS symptoms are: abdominal pain, bloating, satisfaction with stool consistency, epigastric pain, postprandial fullness, early satiety.
Improvement of quality of life assessed through SF-36 questionnaire (eight scale scores) in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients undergoing only a balanced gluten free diet. | 21 days
Improvement of psychological problems and symptoms of psychopathology through the symptom checklist 90 R (SCL 90 R) in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients undergoing only a balanced gluten free diet. | 21 days
Evaluation of the dietary intake in micro and macro-nutrients before and after a Low FODMAP diet or a balanced Gluten Free diet through questionnaire. | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No